CLINICAL TRIAL: NCT05677750
Title: Hematological Disorders Associated With COVID-19 Infection
Acronym: HEMATOCOVID
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Ali Abdelfatah Ahmed, Lecturer, Assiut University
Other Study IDs: 17300633
Record Dates: First submitted 2023-01-06; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hematological Condition With COVID19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed aplastic anemia, ITP, AIHA, Evan syndrome: 40 patients with newly diagnosed aplastic anemia, ITP, AIHA, Evan syndrome. aged one year and older attending Pediatric Hematology Unit at Children University Hospital in Assiut Univesity will undergo the following:
  1. History& Physical Examination:
     History and physical findings will be recorded on a standard data collection sheet.
  2. Bone marrow aspirate and biopsy:
  3. CD 55, CD 59 Flowcytometric markers:
  4. PCR for COVID-19& Antibody for COVID-19
  5. Biologic (Lab) tests:
  Venous blood samples were obtained for:
  * CBC with reticulocytic count and differential
  * Platelet lymphocyte ratio&neutrophil lymphocyte ratio
  * Coagulation profile with PT, PC, INR, PTT
  * Inflammatory markers(ESR,CRP)
  * Serum ferritin, fibrinogin, D-dimer,.

SUMMARY:
The emergence of the Coronavirus Disease -19 (COVID-19) pandemic, has had a tremendous global impact, resulting in substantial morbidity and mortality worldwide.

Although involvement of the lower respiratory track accounts for most of the morbidity and mortality seen, the virus involves several organ systems and the syndrome exhibits clinical diversity with a wide range of symptoms and manifestations.

Aim of this study is to evaluate if there is a casual relationship between the development of aplastic anemias& other immune cytopenias, and recent COVID-19 infection.

DETAILED DESCRIPTION:
Viruses are a form of life that possess genes but do not have a cellular structure. Viruses do not have their own metabolism, and they require a host cell to make new products; therefore, they cannot naturally reproduce outside a host cell (1).

From the hematologist point of view, viruses can play a major role in four conditions: causing infections; causing lymphoproliferations and/or malignancies; causing (pan)cytopenia; and used as vectors in treatment (e.g., gene therapy, CAR-T cells)(2).

Taking into the role of viruses in hematology, pancytopenia, aplastic anemia, and other immune-mediated cytopenias are reported to be related to HIV, Hepatitis viruses, Dengue virus; respiratory infections (community-acquired respiratory virus infections; CARV) caused by Orthomyxoviruses (e.g., influenza A/B), Paramyxoviruses (e.g., human parainfluenza virus PIV-1, -2, -3, and -4; respiratory syncytial virus RSV-A and -B), Picornaviruses (e.g., human rhinovirus), coronaviruses (e.g., human coronavirus), Pneumoviridiae (e.g., human metapneumovirus), and potentially other viruses. (2) A new type of Coronavirus was identified by Chinese authorities in mid-December 2019, named by the Coronavirus Study Group of the International Commission on Virus Classification as "Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)" and the disease was named by the World Health Organization (WHO) as coronavirus disease-2019 (COVID-19). The new virus quickly spread around the world, being declared a pandemic in March 2020.(3) The published data have focused on severe respiratory manifestations, found predominantly in adults, while in children the clinical manifestations are mostly asymptomatic and mild. When the disease is more severe in children, it occurs more frequently in those with less than one year of age or with pre-existing illnesses.(4) Hematological changes are frequent in the COVID-19 disease, such as early lymphopenia and, as the disease progresses, anemia and neutrophilia.(5) Thrombocytopenia can occur secondary to sepsis, disseminated intravascular coagulation or drug-induced,(5) as well as direct bone marrow suppression or immune-mediated destruction.(6)

ELIGIBILITY:
Inclusion Criteria:

* At least one year and less than or equal to 18 years of age
* Newly Diagnosed aplastic anemia, ITP, Autoimmune hemolytic anemia, or Evan syndrome
* Written consent according to institutional guidelines

Exclusion Criteria:

* Hepatitis-associated aplastic anemia (HAAA)
* megaloblastic anemia, bone marrow infiltration (by various cancers or myelofibrosis), and myelodysplastic syndrome or
* acute leukemia.
* Constitutional aplastic anemia
* Any inherited cytopenias
* No written consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 40 patients with newly diagnosed aplastic anemia, ITP, AIHA, Evan syndrome. aged one year and older attending Pediatric Hematology Unit at Children University Hospital
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Complete hematological profile | 12 month
  1. CBC
  2. liver function test
  3. renal chemistry
  4. Coomb's test
  5. serum ferritin
  6. D-dimmer
  7. C reactive protein
Bone marrow aspirate& biopsy: | 12 month
  to detect BM Cellularity
CD55, CD59 flowcytometry | 12 month
  to exclude PNH
PCR &Ab titre for COVID-19 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mai AA Ahmed, MD, Study Director — Assiut University; Mervat A Amin, MD, Principal Investigator — Assiut University; Mustafa M Embaby, MD, Study Chair — Assiut University; Khalid E Elsayh, MD, Study Chair — Assiut University; Dalia T Kamel, MD, Study Chair — Assiut University; Ebtisam SA Hassanin, MD, Study Chair — Assiut University; Hyam Hassan, MD, Study Chair — Assiut University
Locations (1):
- Facility of medicine, Asyut, Egypt